CLINICAL TRIAL: NCT06363825
Title: Single-arm, Prospective Clinical Study of TAE+HAIC Combined With Camrelizumab and Apatinib in the Treatment of Advanced Hepatocellular Carcinoma With High Tumor Load
Brief Title: A Study of TAE+HAIC Combined With Camrelizumab and Apatinib in the Treatment of Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Yiping Chen, Associate professor, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRCTA,ECFAH Of FMU[2024]373
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; high tumor load; camrelizumab; apatinib; HAIC; TAE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): TAE+HAIC combined with camrelizumab and apatinib
  Interventions: Drug: camrelizumab

INTERVENTIONS:
Drug: camrelizumab — TAE: 3-15ml iodized oil;
  HAIC: Indurating arterial catheter, oxaliplatin 85mg/m^2 D1, arterial infusion, lasting 1-2 hours (d1), LV 400mg/m^2, arterial infusion, lasting 2-3 hours (d1), 5-Fu 400mg/m^2, arterial infusion, lasting 3 hours (d1), and fluorouracil 2400 mg/m^2 for 24-48h;
  camrelizumab: 200mg, ivgtt, 30 min (not less than 20 min, not more than 60 min) every 3 weeks (21 days);
  apatinib mesylate: 250mg, once a day, taken orally (the time of daily administration should be as much as possible), with warm water.Stop for 3 days before next cycle intervention.
  Camrelizumab was given intravenously 1 day before TAE+HAIC treatment for each cycle, TAE+HAIC treatment was given on the second day, and oral apatinib was started after discharge.
  Other Names: apatinib

SUMMARY:
To evaluate the efficacy and safety of TAE+HAIC combined with camrelizumab and apatinib in the treatment of advanced liver cancer with high tumor load

DETAILED DESCRIPTION:
At present, there are no prospective clinical studies using the combination regimen (TAE+HAIC+ Apatinib + camrelizumab) in the treatment of advanced liver cancer. Therefore, in this study, investigators designed a single-arm, prospective, multicenter, phase Ⅱ clinical study of arterial infusion of TAE+HAIC+ Apatinib + camrelizumab in the treatment of advanced liver cancer with high tumor load, to explore the safety and efficacy of this regimen. If study gets positive results, it will provide a reference for the subsequent phase Ⅲ clinical trial design, which is expected to provide a new effective approach for the treatment of advanced liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subjects voluntarily joined the study, had good compliance, cooperated with follow-up, and obtained written informed consent;
* 2. Age: 18 years old ≤80 years old, both male and female;
* 3. In accordance with the "Norms for the Diagnosis and Treatment of Primary Liver Cancer (2022 edition)" formulated by the National Health Commission and the 2018 EASL liver Cancer guidelines formulated by the European Association for the Study of Hepatology, a definite diagnosis of hepatocellular carcinoma has been made and pathological results have been obtained;
* 4. There is at least one measurable lesion (spiral CT scan diameter ≥10mm or malignant lymph node short diameter ≥15mm according to RECIST1.1 standard, see Annex 5 for RECIST version 1.1);
* 5. Have not received systematic treatment before;
* 6.CNLC was divided into stages Ⅱa-Ⅲb;
* 7. Meet the status of high tumor load, and meet one of the following conditions: 1) High tumor load is defined according to the 7-11 criteria: combined with the number of tumors and the maximum tumor size, high tumor load is defined as and > 11; 2) Combined with primary branch of portal vein and main cancer thrombus;
* 8. The Child-Pugh classification of liver function is grade A or B (5-8 points);
* 9.ECOG PS score 0-1;
* 10. Expected survival ≥12 weeks;
* 11. If the patient has active hepatitis B virus (HBV) infection: if HBV-DNA≤2000, treatment can be started directly; If HBV-DNA > 2000, start antiviral therapy for one week and then start treatment.
* 12. The major organs function properly and meet the following criteria:

  1. The standard of blood routine examination must meet: (no blood transfusion within 14 days)

     1. Hemoglobin (HB) ≥100g/L,
     2. White blood cell count (WBC)≥3×10^9/L
     3. Absolute neutrophil count (ANC)≥1.5×10^9/L,
     4. Platelet (PLT)≥50×10^9/L;
  2. Biochemical examination shall meet the following standards:

     1. Bilirubin (BIL)<1.5 times the upper limit of normal (ULN);
     2. Alanine aminotransferase (ALT) and aspartate aminotransferase AST<5ULN;
     3. Serum creatinine (Cr) ≤1.5ULN
* 13. Women of childbearing age must have a negative pregnancy test (serum) or urine HCG test within 7 days prior to admission and be willing to use an appropriate method of contraception during the trial period and 8 weeks after the last dose of the test drug; For men, they should be surgically sterilized or consent to an appropriate method of contraception during the trial and for 8 weeks after the last dose of the trial drug.

Exclusion Criteria:

* 1. Pregnant or lactating women;
* 2. Patients with autoimmune diseases, organ/hematopoietic stem cell transplantation, or other malignancies (except cured skin basal cell carcinoma and cervical carcinoma in situ);
* 3. Patients with consciousness disorder or inability to cooperate with treatment, combined with mental illness;
* 4. Patients who have participated in other clinical trials in the past three months;
* 5. Received local treatment (such as surgical resection, radiation therapy, ablative therapy, interventional therapy, etc.) within the past 1 month;
* 6. Thrombotic or embolic events, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism, except portal vein thrombosis, occurred within 6 months prior to the first dose of the study drug;
* 7. Immunosuppressants or systemic hormone therapy (dose >10mg/ day prednisone or other therapeutic hormones) were used within 14 days before enrollment to achieve immunosuppression;
* 8. Esophageal (fundus) varices rupture and bleeding within 1 month before treatment;
* 9. Uncorrectable coagulation dysfunction and severe blood abnormalities, with a tendency to severe bleeding; Platelet count < 50×109/L and severe coagulation dysfunction can not withstand surgery (anticoagulant therapy and/or anticoagulant drug use should be stopped more than 1 week before radiotherapy);
* 10. Refractory ascites, bad fluid;
* 11. Active infection, especially inflammation of the biliary system;
* 12. Severe liver, kidney, heart, lung, brain and other major organ failure;
* 13. Previous use of targeted drugs, any component of PD-1 MAB or other similar tests A quick person;
* 14. Patients with hypertension who cannot be reduced to the normal range by antihypertensive medication (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
* 15. Previous serious cardiovascular disease, including but not limited to the following diseases: Grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥450 ms in men and ≥470 ms in women); According to NYHA criteria, patients with grade Ⅲ to Ⅳ cardiac insufficiency or left ventricular ejection fraction (LVEF) < 50% indicated by cardiac color ultrasound;
* 16. Patients with positive urinary protein (urinary protein test 2+ or more, or 24-hour urinary protein quantity > 1.0g);
* 17. Inability to swallow tablets, malabsorption syndrome or any condition affecting gastrointestinal absorption;
* 18. Patients with other concomitant diseases that, in the judgment of the investigator, endanger the patient's safety or interfere with the patient's completion of the study.
* 19. Patients who do not wish to undergo histological examination to confirm the diagnosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-04-11 (Estimated); Study Completion 2027-05-11 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 years
  Refers to the proportion of all subjects with a best overall result (BOR) of complete remission (CR) or partial remission (PR) as rated according to RECIST 1.1 criteria. If efficacy of CR or PR is achieved, subjects must be confirmed not less than 4 weeks ± 7 days after the initial evaluation.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 1 years
  Refers to the proportion of all subjects with a best overall result (BOR) of complete remission (CR), partial remission (PR), and stable disease (SD) as rated according to RECIST 1.1 criteria.
Progression-free survival (PFS) | 1 years
  PFS was defined as the date from which the subject was first given medication to the date when tumor progression (as assessed by the criteria, with or without continued treatment) was first recorded or the date of death from any cause, whichever came first.
Tumor progression time (TTP) | 1 years
  The definition refers to the time from randomization to the objective progression of the tumor, excluding "death."
Overall survival (OS) | 3 years
  Defined as the time between the date of first dose and the death of the subject due to all causes. Subjects who were alive at the last follow-up visit had OS counted as data censored at the time of the last follow-up visit. The OS of subjects who were lost to follow-up was counted as data censored at the time of last confirmed survival prior to the lost follow-up. OS for data censoring was defined as the time from first dose to censoring.
AE | 1 years
  Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Tang, Principal Investigator — Nanping First Hospital of Fujian Province; Yingchun Li, Principal Investigator — Longyan First Hospital, Affiliated to Fujian Medical University; Peishu Huang, Principal Investigator — Shanghai Sixth Hospital Fujian Hospital; Lei Yu, Principal Investigator — Sanming First Hospital
Locations (1):
- Xinhua Chen, Fuzhou, China

IPD SHARING:
Plan to Share IPD: No